CLINICAL TRIAL: NCT00833079
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Design, Multiple-Site Clinical Study to Evaluate the Bioequivalence of Two Tacrolimus 0.1% Topical Ointment Formulations in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Bioequivalence of Two Tacrolimus 0.1% Topical Ointment Formulations in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TACR-0707
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tacrolimus 0.1% Taro (Experimental): Tacrolimus 0.1% manufactured by Taro applied for 14 days
  Interventions: Drug: Tacrolimus 0.1% manufactured by Taro
- Protopic - Tacrolimus 0.1% (Active Comparator): Protopic, Tacrolimus 0.1% applied for 14 days
  Interventions: Drug: Protopic - Tacrolimus 0.1%
- Vehicle (Placebo Comparator): Tacrolimus vehicle applied for 14 days
  Interventions: Drug: Tacrolimus Vehicle manufactured by Taro

INTERVENTIONS:
Drug: Tacrolimus 0.1% manufactured by Taro — Treatment applied as a thin layer to target area twice daily for 14 days
  Arms: Tacrolimus 0.1% Taro
Drug: Protopic - Tacrolimus 0.1% — Treatment applied as a thin layer to target area twice daily for 14 days
  Arms: Protopic - Tacrolimus 0.1%
Drug: Tacrolimus Vehicle manufactured by Taro — Treatment applied as a thin layer to target area twice daily for 14 days
  Arms: Vehicle

SUMMARY:
The primary objectives are to establish the therapeutic equivalence of tacrolimus ointment 0.1%, manufactured by Taro Pharmaceuticals Inc. and Protopic® (tacrolimus), 0.1% topical ointment (Astellas Pharma US, Inc.) and to show superiority over vehicle in the treatment of moderate to severe atopic dermatitis.

The secondary objectives are to compare the adverse event (AE) profiles of the two ointments and to investigate their systemic absorption at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, 18 years of age or older.
* Patient has documented evidence that they have been unresponsive to alternative more traditional therapies such as topical corticosteroids, or in the investigators opinion, such first line therapy would be deemed inadvisable because of potential risks to the patient.
* If female and of child bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, IUD, oral, transdermal, injected or implanted hormonal contraceptives).
* Have confirmed diagnosis of atopic dermatitis using the diagnostic features as described by Hanifin and Rajka.
* Have an IGSA score of 3 (moderate) or 4 (severe)
* Have an affected Body Surface Area (BSA) of at least 20%
* Have a minimum Eczema Area and Severity Index (EASI) score of at least 15

Exclusion Criteria:

* Mild atopic dermatitis as defined by IGSA score of 0 (clear), 1 (almost clear), or 2 (mild) OR %BSA affected less than 20% OR EASI Score of less than 15.
* Clinically infected atopic dermatitis at the baseline visit. Tacrolimus is not indicated for the treatment of clinically infected atopic dermatitis
* Any dermatological condition other than atopic dermatitis that in the Investigator's opinion may interfere with the evaluation of the patient's atopic dermatitis
* Females who are pregnant, lactating or likely to become pregnant during the study.
* History of allergy or sensitivity to tacrolimus, pimecrolimus, any macrolides such as clindamycin erythromycin
* Current diagnosis or history or any disease, which in the Investigators opinion would contraindicate the use of immunosuppressants, including but not limited to human immunodeficiency virus (HIV) and cancer.
* Use of any nonsteroidal immunosuppressants
* Regular use of intranasal or inhaled corticosteroids, greater than the equivalent of 2 mg of prednisone/day, within 14 days of the first dosing day.
* Use of non-sedating histamines are not allowed for at least 7 days prior to the first dosing day or throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
ISGA score 0 or 1 | 14 days

SECONDARY OUTCOMES:
% change in BSA | 14 days
% change in EASI | 14 days
% change in ISGA | 14 days
Safety and adverse event profile | 14 days